CLINICAL TRIAL: NCT00720343
Title: Effect of Oral Choline Supplementation on Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAC8413; 1R21AT004708-01A1 (NIH)
Record Dates: First submitted 2008-07-21; First posted 2008-07-22 (Estimated); Results first posted 2016-03-25 (Estimated); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Postoperative Pain; Inflammation
MeSH Terms: conditions — Pain, Postoperative; Inflammation | interventions — Choline; Gelatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Choline (Experimental): Oral choline
  Interventions: Drug: Choline
- Placebo (Placebo Comparator): Gelatin Capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Choline — Oral Choline 20 grams before surgery
  Other Names: Tricholine 1200
  Arms: Choline
Drug: Placebo — Gelatin Capsule
  Other Names: Gelatin Capsule
  Arms: Placebo

SUMMARY:
This research will test whether consuming additional choline before gynecological surgery decreases postoperative pain.

DETAILED DESCRIPTION:
More than 70% of the patients undergoing surgery in the USA, experience moderate to severe pain after the surgery in spite of being treated for pain. We will test whether choline will produce an effective additional analgesic action for postoperative pain treatment. Choline and lecithin are safe and are available for consumers as over-the-counter nutritional supplements. Choline supplementation decreases postoperative pain in rodents. Also Nicotine decreases postoperative pain in humans and since choline acts on the same receptors as nicotine, choline supplementation may be effective as an analgesic without the risks of addiction and the side effects like high heart rate and blood pressure.

Sixty women between the ages 18 and 60 undergoing open abdominal gynecological surgeries will be studied. We will not study people with chronic pain, drug abuse, and/or nicotine use over the past six months, current pregnancy or breastfeeding, allergy to soy, or inability to take any drug that we will use in the study.

Patients will take 10 tablets (choline or gelatin powder placebo) the night before surgery. After anesthesia, a second dose will be given into a tube that goes into the patient's stomach. One tablespoon of blood (15 mL) will be drawn five times to measure genetics, changes in levels of plasma choline and inflammatory markers: blood will be drawn at the preoperative visit, three times on the day of surgery and once 24 hours postoperatively. At 24 hours after surgery and on their follow-up visit with their doctor, the patient's surgical wound will be photographed and patients will complete a survey on satisfaction with treatment.

Primarily we are looking at the pain scores after surgery and secondarily at the pain medication use, plasma choline levels, wound healing and satisfaction with pain treatment.

This is a randomized double blind study. Patients will consume ten tablets (10g choline or placebo) the night before undergoing gynecological surgery and 10 tablets the morning of surgery. We will measure pain after surgery, baseline and postoperative plasma choline, and test genetics.

ELIGIBILITY:
Inclusion Criteria:

* open pelvic surgery
* able to swallow pills

Exclusion Criteria:

* chronic pain
* opioid use
* pregnancy
* lactation

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Flood, MD, Principal Investigator — Stanford University
Locations (1):
- New York Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sidhu N, Davies S, Nadarajah A, Rivera J, Whittington R, Mercier RJ, Virag L, Wang S, Flood P. Oral choline supplementation for postoperative pain. Br J Anaesth. 2013 Aug;111(2):249-55. doi: 10.1093/bja/aet031. Epub 2013 Apr 7. PMID 23568851

RESULTS

PARTICIPANT FLOW:
Groups:
- Choline: Participants ingested ten tablets (GNC Triple Lecithin 1200 choline tablets) containing 12 g of high choline lecithin and 4.2 g phosphatidyl choline the night before surgery. On the day of surgery, a second dose of study drug (equivalent to ten tablets) was administered by the clinical anesthesiologist as a slurry through the oral gastric tube that was placed after induction of general anesthesia.
- Placebo: Participants ingested ten gelatin capsules the night before surgery. On the day of surgery, a second dose of the placebo (equivalent to ten capsules) was administered by the clinical anesthesiologist as a slurry through the oral gastric tube that was placed after induction of general anesthesia.
Period: Overall Study
Arm/Group | Choline | Placebo
Started | 30 | 30
Completed | 29 | 28
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Choline | Placebo | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Customized [Count of Participants; unit: Participants]
  18-21 years | 0 | 0 | 0
  22-59 years | 29 | 28 | 57
  >60 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 20 | 17 | 37
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 18 | 38
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale (NRS) Pain Score
Description: NRS range is 0-10 where 0 is no pain and 10 is the worst pain imaginable
Time Frame: End of surgery, and 1 hour after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Choline | Placebo
Number analyzed (Participants) | 29 | 28
score on a scale
  End of surgery | 5.8 (2.2) | 7.4 (1.7)
  1 hour after surgery | 7.4 (5.2) | 8.8 (3.2)

2. Secondary Outcome: Amount of Morphine Used by Participants Post-surgery
Time Frame: 1 hour after surgery, and 24 hours after surgery
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | Choline | Placebo
Number analyzed (Participants) | 29 | 28
mg
  1 hour after surgery | 3.6 [1 to 6] | 4 [1 to 8]
  24 hours after surgery | 49 [31 to 71] | 48 [33 to 62]

ADVERSE EVENTS:
Time Frame: Up to 24 hours post-surgery
Arm/Group | Choline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 0/29 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No